CLINICAL TRIAL: NCT05576025
Title: Effects of Cold-induced Shivering at Different Intensities on 24-hour Glucose Profiles in Pre-diabetic Individuals and Patients With Type 2 Diabetes Mellitus
Brief Title: Acute Effects of Cold-induced Shivering on 24-hour the Glucose Profile in Metabolically Compromised Populations
Acronym: SHIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL.81053.068.22; NL.81053.068.22 / METC 22-026 (Registry Identifier: Central Committee on Research Involving Human Subjects)
Record Dates: First submitted 2022-09-26; First posted 2022-10-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus; Pre-diabetes
Keywords: Lifestyle intervention; Cold exposure; Prevention; Treatment; Metabolic health; Glucose homeostasis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: In a randomised cross-over design participants will be exposed to two different intensities of shivering thermogenesis, namely mild and moderate. There will be a wash-out period of at least 3 weeks between the interventions.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1: Shivering intensity 1 (Experimental): During Arm 1 of the study participants will undergo the first cold exposure at either mild or moderate shivering intensity (depending on the randomisation).
  Interventions: Other: Lifestyle intervention (cold exposure)
- Period 2: Shivering intensity 2 (Experimental): During Arm 2 of the study participants will undergo the second cold exposure at the alternative shivering intensity.
  Interventions: Other: Lifestyle intervention (cold exposure)

INTERVENTIONS:
Other: Lifestyle intervention (cold exposure) — Participants will undergo two cold exposures with different shivering intensities. Mild shivering is defined as energy expenditure increased by 1.5-fold compared to the resting metabolic rate. Moderate shivering is 2.5-fold increase in metabolic rate.

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) and its associated comorbidities pose a major health concern worldwide. Although lifestyle strategies, such as exercise and diet-induced weight loss are effective interventions to counteract the development and progression of the disease, its prevalence continues to increase. Therefore, alternative therapeutic strategies are warranted. One such method, which has increasingly been gaining attention, is cold exposure. Previously, investigators have shown that exposing T2DM patients to mild cold (14-16 oC) for 6 hours per day for 10 consecutive days enhanced their insulin sensitivity by ~43%. This remarkable improvement in insulin sensitivity was accompanied by robust GLUT4 translocation in the skeletal muscle of participants, which likely mediated the improvements in insulin-stimulated glucose uptake. Follow-up research suggested that a certain degree of muscle activation/shivering appears to be a prerequisite for the cold-induced enhancement in skeletal muscle insulin-stimulated glucose uptake. In humans however, very little information is available about the effects of shivering on glucose metabolism, especially in metabolically compromised individuals. Therefore, in this study, the aim to investigate the acute effects of (different intensities of) shivering on 24-hour glucose profiles in pre-diabetic individuals as well as in T2DM patients. For that purpose, a focus will be placed on clinically relevant glycaemic parameters by means of continuous glucose monitoring, which is increasingly being used in T2DM management and prevention.

DETAILED DESCRIPTION:
Participants will be recruited in and near the vicinity of Maastricht by advertising on local billboards, in local newspapers, public spaces, contacting previous participants who gave consent to be contacted again, and on the internet. Those who express interest will be invited for a screening. Upon arrival at the research facility, participant will sign an informed consent form (see chapter 11.2 for complete procedure). Subsequently, measurements of height, weight and blood pressure will be performed. The blood pressure measurement will be performed 3 times to obtain an average blood pressure value (to avoid measuring a peak or dip in the pressure). Furthermore, a 10-lead electrocardiogram (ECG) will be recorded and the subjects will fill out a medical history (see document F1.1). Following this, a two-hour oral glucose tolerance test (OGTT) will be performed to assess glucose tolerance (applies only for potential pre-diabetic subjects). Fasting blood sample (19 mL in total) from the T2DM patients will be obtain via venepuncture and no OGTT will be performed. After inclusion in the study, participants will undergo two study periods (period 1 and period 2) of eight days. During each period, participants will visit the research facilities three times.

Sample size:

The primary aim of this study is to determine if acute cold-induced shivering will decrease the area under the curve (AUC) for 24-hour glucose of individuals with a different degree of metabolic impairment, including pre-diabetic participants and patients with T2DM. Thus, the study will be powered accordingly to allow for detecting the expected minimal effect in both groups. It is expected to see a clinically meaningful decrease in AUC for 24-hour glucose of at least 15% in the pre-diabetic participants. Based on literature, investigators anticipate a more pronounced (20%) effect in 24-hour AUC for glucose in T2DM patients. To ensure that both groups are powered appropriately, the sample size calculation of the T2DM patients will be followed and 12 participants will be included in each group. When a drop-out rate of 20% is considered, investigators anticipate that up to 15 participants will need to be included in each group to reach this sample size. From experience with similar studies it is estimated that there will be a screening failure of 50% and 70% for the T2DM and pre-diabetes groups, respectively. Therefore, it is expected that researchers will need to screen 30 and 50 individuals, respectively, from each study population.

Use of co-interventions: to minimise the variability in blood glucose induced by diet, all participants will be asked to consume standardised meals during the two study periods. Additionally, subjects will be asked to avoid strenuous physical activity (e.g. walking long distances, stair climbing for >10 minutes or cycling for >30 min, hiking) or structured exercise during the study periods to minimize exercise induced variability in blood glucose. In addition, participants are asked to withstand from alcohol and caffeine-containing drinks 24 hours before and after cold exposure. Participants will be instructed to keep their normal sleeping pattern throughout the entire study. During wash-out participants are advised to maintain their normal dietary habits and activity pattern.

Measurements:

Participants will be equipped with a continuous glucose monitor (CGM) to continuously measure blood glucose during each study period. Participants will be asked to wear a FreeStyle Libre Pro iQ (Abbott) glucose monitor, which is a system able to measure reliable blood glucose levels over a longer period; it is a standard technique in daily diabetes practice. To determine physical activity levels throughout both study periods, participants will be asked to wear an activPAL activity monitor (PAL Technologies Ltd). Respiratory gas exchange will be measured using an open-air circuit respirometry with an automated ventilated hood system (Omnical, Maastricht Instruments, Maastricht University, Maastricht, The Netherlands). The O2 (oxygen) consumption and CO2 (carbondioxide) production will be measured, from which energy expenditure and substrate oxidation can be calculated. Core temperature will be measured during the two cold exposure interventions with a telemetric pill (BodyCap, France) that will be swallowed in the evening before each cold exposure day. During the two cold exposure days (visit 2 and 5) surface electromyography (EMG) sensors (Trigno wireless system, Delsys Inc., USA) will be attached to the surface of 6 muscles (upper trapezius fibres, latissimus dorsi, pectoralis major, vastus lateralis, vastus medialis, rectus femoris) to determine skeletal muscle electrical activity. Prior to the start of the cold exposure intervention during visit 2 and 5 a catheter will be inserted in the antecubital vein of the participant to repeatedly draw blood during the intervention. Blood samples will be collected in the appropriate tubes and immediately centrifuged at high speed and plasma will be immediately frozen in liquid nitrogen and stored at -80 ̊C for later analysis. Blood will be analyzed for: glucose, insulin, cholesterol, triglycerides, free fatty acids and other relevant metabolic health markers. Subjects will be provided with standardised meals for both study periods (same period as the CGM measurements are performed). The total daily caloric intake will be determined by multiplying the basal metabolic rate (BMR) of the subject by a PAL value, where the BMR will be estimates using the Harris-Benedict formula. Since our participants are sedentary by study design, a PAL value of 1.5 for participants aged <50 years and 1.4 for subject aged 50-75 will be used, as done in a previous study within the same research group (NL78281.068.21). The caloric distribution throughout the day and the macronutrient composition of the meals will maximally reflect the habitual diet of the Dutch population. As such, the breakfast, lunch and dinner will account for ~20-25%, ~20-25% and ~40-45% of the total caloric intake, respectively, and snacks will account for up to 10%.

Statistical analysis:

For all study parameters data will be reported as minimum, maximum, mean ± SD and/or ± SEM, or as median and range in case of a highly skewed distribution. All primary, secondary, and explorative study parameters are numerical values or an average of numerical values of a defined time period. Statistical analyses will be performed using the statistical computer program SPSS version 26.0. P-values of ≤ 0.05 (two-sided testing) will be considered statistically significant. Missing values will not be replaced. If a missing value occurs for a specific parameter, the subject in question will not contribute to the analysis of that parameter and therefore no intention-to-treat procedure will be followed but a per protocol analysis. Only participants who fully complied with the study protocol and fulfilled the entire study will be included in the analysis of the outcome parameters. Paired sample t-test analysis will be conducted to investigate the effects of shivering on the primary outcome (24-hour AUC for glucose measured before vs. after acute shivering) in the two study groups. The secondary outcome (24-hour AUC for glucose in response to acute mild vs. moderate shivering) will be investigated using a linear mixed model with treatment (shivering intensity) and time as fixed factors.

Safety reporting:

In accordance to section 10, subsection 4, of the WMO, the sponsor will suspend the study if there is sufficient ground that continuation of the study will jeopardise subject health or safety. The sponsor will notify the accredited METC (Medical Ethics Commitee) without undue delay of a temporary halt including the reason for such an action. The study will be suspended pending a further positive decision by the accredited METC. The investigator will take care that all subjects are kept informed.

Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the cold exposure intervention/trial procedure. All adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded.

The investigator will report all (Serious Adverse Events) SAEs to the sponsor without undue delay after obtaining knowledge of the events.

The sponsor will report the SAEs through the web portal ToetsingOnline to the accredited METC that approved the protocol, within 7 days of first knowledge for SAEs that result in death or are life threatening followed by a period of maximum of 8 days to complete the initial preliminary report. All other SAEs will be reported within a period of maximum 15 days after the sponsor has first knowledge of the serious adverse events.

Data monitoring:

The study will be monitored by the Clinical Trails Centre Maastricht (CTCM). The study is classified as a clinical trial with negligible. In accordance with this risk classification, in total, three monitor visits will be performed: initial, interim and close out visit. During these visits source data verification (including electronic case report forms, medical records, etc.) and overall quality assurance will be performed by the accredited monitor.

The sponsor/investigator will submit a summary of the progress of the trial to the accredited METC once a year. Information will be provided on the date of inclusion of the first subject, numbers of subjects included and numbers of subjects that have completed the trial, serious adverse events/ serious adverse reactions, other problems, and amendments.

The investigator/sponsor will notify the accredited METC of the end of the study within a period of 8 weeks. The end of the study is defined as the last patient's last visit. The sponsor will notify the METC immediately of a temporary halt of the study, including the reason of such an action.

Handling and storage of data and documents:

At the start of the study, participants will be assigned a study code (SHVR + number of inclusion) that will not change during the study. The code will consist of the study acronym and a number in sequential order of screening; i.e. SHVR001, SHVR002, SHVR003, etc. This code will be followed with the period, P1 or P2. This code is linked with the name, address, date of birth, and telephone number of the participant in a password protected file. For all purposes, this code will be used for participant identification. Only the responsible principal investigator (Joris Hoeks) and the researcher conducting this study (Dzhansel Hashim) can access this file. The privacy of the participants who take part in the study will be protected. This means that the study code will not contain the participants' initials or birth date as explained above. In case data, documents or samples will be analyzed outside the scope of this proposed study, the participants will be asked for permission but only if the participant provided permission to be approached for follow-up research on the informed consent. Data files containing personal information of participants are stored separately and password protected. All human material, research data and documents will be stored for 15 years.

Ethical consideration:

This study will be conducted according to the principles of the Declaration of Helsinki (64th WMA General Assembly, Fortaleza, Brazil, October 2013) and in accordance with the Medical Research Involving Human Subjects Act (WMO) and other guidelines, regulations and Acts.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all subjects:

* to be able to provide signed and dated written informed consent prior to any study specific procedures
* have suitable veins for cannulation or repeated venepuncture
* male, or postmenopausal (at least 1 year post cessation of menses) female
* aged 40 - 75 years
* have stable dietary habits (no weight loss or gain >5 kg within the past 3 months)
* have no signs of active cardiovascular disease or liver malfunction
* have body mass index (BMI) >= 27 and <= 38 kg/m2

Additional inclusion criteria for pre-diabetic subjects:

Pre-diabetes based on one or a combination of the following criteria:

* Impaired Glucose Tolerance (IGT): plasma glucose values ≥ 7.8 mmol/l and ≤ 11.1 mmol/l 120 minutes after glucose drink consumption during OGTT in screening
* ImpairedFastingGlucose(IFG):Fastingplasmaglucose≥6.1mmol/land≤6.9 mmol/l
* Insulin Resistance: glucose clearance rate ≤ 360 mL/kg/min, as determined using OGIS120
* HbA1c of 5.7-6.4%

Additional inclusion criteria for type 2 Diabetes Mellitus patients:

* being diagnosed with T2DM at least 1.5 years before the start of the study
* have well-controlled diabetes, i.e. HbA1c levels < 8.5%
* have no signs of active diabetes-related co-morbidities, including active cardiovascular diseases, diabetic foot, polyneuropathy or retinopathy
* diet treatment OR on an oral glucose lowering medication: metformin only or in combination with sulfonylurea agents and/or on stable dose of a DPPIV inhibitor treatment for at least the last 3 months

Exclusion Criteria:

* not meeting the respective inclusion criteria
* participation in a clinical study with an investigational product during the last 3 months or as judged by the investigator
* uncontrolled hypertension
* having Hb <8 mmol/L (men), Hb <7 mmol/l (women)
* consuming alcohol >2 servings per day (man) or >1 servings per day (women)
* not wanting to be informed about unexpected medical findings during the screening
* being engaged in structured exercise > 2h per week
* smoking
* being cold-acclimated, e.g. having taken daily extended cold baths, working in a refrigerated environment, or practicing regular cold-water swimming/showering within 1 month of starting the study

Exclusion criteria specific for pre-diabetic subjects:

- Type 2 Diabetes Mellitus

Exclusion criteria specific for type 2 Diabetes Mellitus patients:

- being insulin-dependent and/or using SGLT2 inhibitor medications

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
24-hour area under the curve (AUC) for glucose | 24-hour period before and after each shivering session
  24-hour AUC for glucose expressed in mmol/L x min

OTHER OUTCOMES:
Average 24-hour interstitial glucose concentration | 24-hour period before and after cold exposures and 72-hour periods before/after cold exposures
  Measured in mmol/L
Time above range (TAR) | Over a period of 72 hours before and after the two cold exposures
  Measured in minutes; reflects the total duration for which glucose concentration was above the normal physiological levels
Glucose variability | 72-hour period before and after each cold exposure and following each meal
  Measured in % coefficient of variation; reflects how dynamic the changes in blood glucose levels are over a period of time
Energy expenditure during shivering | Over a period of 3-4 hours during each cold exposure
  Average energy expenditure expressed in kJ/min
Substrate oxidation | Over a period of 3-4 hours during each cold exposure
  Oxidation of carbohydrate and fat during cold exposure, expressed in g/min
Sedentary time | Over the 96 and 72-hour period before and after each cold exposure, respectively
  Expressed in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joris Hoeks, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Department of Nutrition and Movement Sciences, Maastricht, Limburg, Netherlands